CLINICAL TRIAL: NCT06031051
Title: Capsule Endoscopy as an Alternative to Colonoscopy. Could the Number of Colonoscopies be Reduced?
Brief Title: Capsule Endoscopy as an Alternative to Colonoscopy
Acronym: CAPSUCOVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Begoña González Suárez, MD PhD, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAPSUCOVID
Record Dates: First submitted 2023-03-01; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Colonic Disease
MeSH Terms: conditions — Colonic Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pillcam Crohn's Capsule Endoscopy and colonoscopy (Other): All patients will be submitted to a Pillcam Crohn's Capsule Endoscopy (Medtronic) previous their colonoscopy
  Interventions: Device: Pillcam Crohn's Capsule Endoscopy

INTERVENTIONS:
Device: Pillcam Crohn's Capsule Endoscopy — Patients with scheduled colonoscopy are invited to a previous exploration with capsule endoscopy
  Other Names: Pillcam

SUMMARY:
This is a prospective, multicenter, interventional study assessing CE, in patients already scheduled for colonoscopy at tertiary referral hospitals, as a technique to reduce the number of unnecessary colonoscopies and identify patients to prioritize in endoscopy waiting lists.

DETAILED DESCRIPTION:
Study design Enrolled patients already scheduled for non-urgent colonoscopy according to local practice will be offered to undergo an early CE; in case of negative proof they will perform colonoscopy as already planned (scheduled colonoscopy); in patients with positive findings, requiring endoscopic treatment or intervention, colonoscopy will be performed within 30 days from CE (early colonoscopy).

Study population Patients who received the indication for colonoscopy as per clinical practice and subsequently identified as non-urgent procedures, according to locally established prioritization criteria

ELIGIBILITY:
Inclusion Criteria:

* Iron deficiency anaemia with or without a colonoscopy performed within the last 5 years

  * Rectal bleeding/haematochezia in patients >50 years who have undergone a colonoscopy <5 years ago or <50 years with no risk factors for CRC
  * Chronic constipation/abdominal distension/abdominal pain/diarrhea
  * Suspected CRC due to clinical criteria (NICE guidelines 2015, updated in 2017) with no iFOBT performed
  * Recent change in bowel habits
  * Follow-ups: post-polypectomy syndrome, family history of CRC, hereditary syndromes, CRC surgery, Inflammatory Bowel Disease

Exclusion Criteria:

* Study following an episode of complicated acute diverticulitis or with an uncertain diagnosis of acute diverticulitis
* Evaluation following fragmented resection (recurrence ruled out)
* Patients with a positive FIT
* Pregnancy or breast-feeding
* Any contraindication to Crohn's Capsule endoscopy such as known or suspected gastrointestinal obstruction, strictures or fistulas, a previous altered Patency capsule, dysphagia or other swallowing disorders and cardiac pacemakers or other implanted electromedical devices.
* Allergy or known contraindication to the medications and preparations agents used in the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
percentage of patients who could avoid colonoscopy | 6 months
  To evaluate the percentage of patients who could avoid colonoscopy by performing a previous CE

SECONDARY OUTCOMES:
CE diagnostic yield and adenoma detection rate (ADR) | 6 months
  Number of adenoma detected by CE
To compare CE and CC findings | 6 months
  Compare findings between both techniques

CONTACTS AND LOCATIONS:
Overall Officials: BEGOÑA GONZALEZ SUAREZ, MD PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital universitario de Santa Cruz de Tenerife, Santa Cruz de Tenerife, Canary Islands
  - Hospital clinic of barcelona, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Mutua de Terrassa, Terrassa

IPD SHARING:
Plan to Share IPD: No